CLINICAL TRIAL: NCT05727696
Title: A Comparative Study Between Radius and Capitate Shortening in Ulna Minus Variance Kienbock's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alamir Mohamed Farrag, residant orthopedic departement, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: soh-med-23-01-10
Record Dates: First submitted 2023-02-05; First posted 2023-02-14 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Avascular Necrosis of Lunate
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radial shortening (Active Comparator)
  Interventions: Procedure: Henry approach; volar approach
- capitate shortening (Active Comparator)
  Interventions: Procedure: dorsal approach

INTERVENTIONS:
Procedure: Henry approach; volar approach — Radial Shortening : Supine position, general anesthesia, volar approach, Henry approach, osteotomy 1 inch from radio-carpal joint surface, shortening 2.5 mm of distal shaft radius, fixation by small DCP or small T plate.
  Arms: radial shortening
Procedure: dorsal approach — Capitate Shortening : Supine position, general anesthesia, dorsal approach, separation between 2nd and 3rd compartments of extensor tendons, osteotomy & shortening 2.5 mm of capitate, compression by Herpert screw.
  Arms: capitate shortening

SUMMARY:
1. Kienböck's disease refers to avascular necrosis of the lunate carpal bone, known as lunatomalacia. It was first recognized and described by Austrian radiologist Robert Kienböck's in 1910
2. The lunate is the central bone in the proximal row, and it articulates with the scaphoid, capitate, triquetrum, and occasionally the hamate. More proximally, the lunate is a component of the radiocarpal joint, and it also articulates with the ulna via the triangular fibrocartilage complex (TFCC)
3. The exact cause of Kienböck's is not known, though there are thought to be a number of factors predisposing a person to Kienböck's. Although there is no evidence that Kienböck's disease is inherited, it is possible that unidentified genetic factors could contribute to the development of the condition, It is multifactorial, related to the following variables:Ulnar negative variance (or ulna minus),Vascular supply to the lunate bone,Lunatemorphology,Radial inclination angle,multiple wrist trauma
4. Kienböck's disease is the second most common type of avascular necrosis of the carpal bones, preceded only by avascular necrosis of the scaphoid. The typically affected population is males aged 20-40 years
5. Patients usually present with unilateral pain over the dorsal aspect of the wrist, limited wrist motion, weakness, or a combination of the three. Wrist extension and axial loading exacerbate pain. Symptoms range from mild to debilitating. It is rarely bilateral, and trauma is often absent. Physical examination commonly reveals wrist swelling, tenderness over the expected location of the lunate, synovitis, and loss of grip strength
6. Kienböck's disease is a clinical and imaging diagnosis. Both radiography/computed tomography and magnetic resonance imaging (MRI) are highly specific. However, MRI is the most sensitive and detects radiographically occult cases

ELIGIBILITY:
Inclusion Criteria:

* Age : 18-65 Years.
* Stages II & III.
* Ulna minus.

Exclusion Criteria:

* Teens.
* Serious medical condition.
* Stage I& IV.
* Sever osteoporosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
(Modified Mayo Wrist Score) | 1 year
  wrist pain ; hand grip; work status ; range of motion

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided